CLINICAL TRIAL: NCT04394078
Title: Impact of COVID-19 Pandemic on Depression and Quality of Life: Cross Sectional Study on Turkish Society and Suggestions on Potential Solution
Brief Title: Impact of COVID-19 Pandemic on Depression and Quality of Life
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Begüm Okudan, MSc. Pt, Okan University
Other Study IDs: 56665618-204.01.07
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Depression; Quality of Life; Covid 19; Social Isolation
Keywords: Covid 19; Depression; Quality of Life; Turkish Society; Social Isolation
MeSH Terms: conditions — Depression; COVID-19; Social Isolation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Turkish society: Individuals speak Turkish and lives in Turkey, ages between 15 - 65, literate and with internet access
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Volunteer individuals enrolled the study after approval an online informed consent form. Sociodemographic data of the participants recorded as an online survey. Then, patient reported outcomes were used to assess depression (Zung depression Scale) and quality of life (WHO Qualiy of Life - Bref version).

SUMMARY:
It is aimed to investigate the depression and quality of life of Turkish society caused by Covid-19 pandemic and reveal the relationship between them

DETAILED DESCRIPTION:
Study hypothesis that people are tend to be depressed and the quality of life is affected negatively by Covid-19 pandemic. Although Turkey has affected moderately, the immediate change on depression and quality of life observable and measurable. It is aimed to investigate the depression and quality of life of Turkish society caused by Covid-19 pandemic and reveal the relationship between them. According to existing data and perspective of psychology and physiotherapy, potential solutions will be aligned.

ELIGIBILITY:
Inclusion Criteria:

* being Turkish
* understanding Turkish
* currently living in Turkey
* being between the age of 15 - 65
* being literate
* have internet access

Exclusion Criteria:

* being diagnosed with a psychological disorder before the pandemic
* having missing value on outcome measures
* giving incomprehensible answering

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of the individuals between 15 - 65 ages in Turkey is 56.391.925 people. It is calculated that there are 42.463.119 individuals cover the criterion as universe of the study.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Sociodemographic information form | two months after Covid 19 recognised as pandemic
  Participants are asked to give information about: age, gender, educational status, height, weight, occupation, working status, city inhabited, whether they live alone or with someone, whether they have a chronic disease, have a pet, do physical activity, eat healthy and sufficient, have qualified sleep, whether they are supported economically.
Zung Depression Scale | two months after Covid 19 recognised as pandemic
  Zung depression scale, developed by Zung (Zung, 1965), is patient rating depression scale, was used to asses four domains related to depression; somatic, mood disorders, psychomotor and psychological disorders. Each question is rated on a 4-point Likert scale (0- never, 1- sometimes, 2- frequently, 3- always). Scale contains 10 straight 10 reverse questions. The total score is calculated from the raw score obtained (total score = (raw score / 80) * 100). Accordingly, scores less than 50 are normal or no psychopathology; between 50 and 59 points indicates mild level, between 60 and 69 points indicate moderate level and 70 and above points indicate severe level depression (Thurber et al., 2002). The validity reliability of the scale was studied on Turkish society (Gencdogan & Nihal, 2011)
World Health Organization Quality of Life - Bref | two months after Covid 19 recognised as pandemic
  World Health Organization Quality of Life Bref is the short version of the WHOQOL-100 to assess the health-related quality of life (Harper et al., 1998), which has efficient psychometric properties, valid and reliable for Turkish society (Eser et al., 1999). It is essential for epidemiological survey and international report has built for psychometric properties for 26 country where Turkey within (Skevington et al., 2004). It has 4 domains; physical health, psychology, social relations and environment. Each question is answered on a 5-point Likert scale. The raw score is converted into a percentage system. The quality of life is interpreted as good as it gets closer to 100% (Akvardar et al., 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data are stored by researches, if needed for scientific purposes, it can be discussed to share .